CLINICAL TRIAL: NCT07225010
Title: Fostering Healthy Relationships Through Tele-PCIT for Families of South Carolina
Brief Title: Tele-PCIT for Healthy Relationships in Families At-Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Principal Investigator, Rosmary Ros-Demarize, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00146035; 2167-SP (Other Grant/Funding Number: Duke Endowment)
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Disruptive Behavior; Pediatrics
MeSH Terms: conditions — Problem Behavior | interventions — RTI 121

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-PCIT (Experimental): Families in the Tele-PCIT condition will recieve a time limited (10 session) version of PCIT via telehealth.
  Interventions: Behavioral: Telehealth Parent Child Interaction Therapy
- Waitlist Control (Other): Delayed Start of Tele-PCIT
  Interventions: Behavioral: Telehealth Parent Child Interaction Therapy (Delayed Start)

INTERVENTIONS:
Behavioral: Telehealth Parent Child Interaction Therapy — During tele-PCIT, therapists coach parents on parenting strategies while they play with their child during one hour weekly sessions. The first phase of therapy focuses on increasing positive behaviors and the second phase focuses on decreasing negative behaviors with discipline strategies. The therapist and the family will be connected through a video feed on either a phone, tablet, or computer and a Bluetooth headset.
  Other Names: Tele-PCIT; iPCIT
  Arms: Tele-PCIT
Behavioral: Telehealth Parent Child Interaction Therapy (Delayed Start) — Delayed start of 12-weeks for delivery of Tele-PCIT. During tele-PCIT, therapists coach parents on parenting strategies while they play with their child during one hour weekly sessions. The first phase of therapy focuses on increasing positive behaviors and the second phase focuses on decreasing negative behaviors with discipline strategies. The therapist and the family will be connected through a video feed on either a phone, tablet, or computer and a Bluetooth headset.
  Other Names: Tele-PCIT; iPCIT
  Arms: Waitlist Control

SUMMARY:
The study will examine Parent Child Interaction Therapy (PCIT) delivered via telehealth (Tele-PCIT) for young children at risk for adverse childhood experiences and/or trauma exposure.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the feasibility, acceptability, engagement, and initial efficacy of time-limited Parent Child Interaction Therapy (PCIT) delivered via telehealth (Tele-PCIT) across 40 young children at risk for adverse childhood experiences and/or trauma exposure. The study compares outcomes between families receiving Tele-PCIT (n = 20) and those assigned to a waitlist control (n = 20). All families will complete baseline, post, and follow-up evaluations to assess child behavioral outcomes, parenting outcomes, and trauma symptoms. In order to be eligible children are between 2 and 7 years of age presenting with behavioral concerns and scoring at-risk on childhood averse events measures.

ELIGIBILITY:
Inclusion Criteria:

* Child participants must:

  * Be between 2:0-6:11 years old
  * Have elevated levels of disruptive behavior problems as defined by the Eyberg Child Behavior Inventory (ECBI)
  * Have receptive language appropriate for PCIT (approximately 2-years old)
  * Medicaid eligible, or be uninsured
  * Score of 1 or greater on an ACEs (adverse childhood experiences) measure (PEARLS)
* Parent participants must:

  * Be the child's legal guardian
  * Be able to provide consent for themselves (i.e., have decision making capacity and do not need a legally authorized representative themselves).
  * Must be living with the child

Exclusion Criteria:

* None

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Parenting Practices | Assessed at Baseline, 12-weeks post baseline, and at a 3-month follow-up
  Measured by the Parenting Scale. The parenting scale is comprised of 30 items rated 1-7 with specific items being averaged to create composites for Laxness, Verbosity, and Overreactivity. Higher scores on each scale indicate higher levels of each parenting behavior.
Child Behavior | Assessed at Baseline, 12-weeks post baseline, and at a 3-month follow-up
  Measured by Eyberg Child Behavior Inventory. The ECBI is comprised of 36 items ranging from 1 to 7 and the overall score has a a minimum of 36 and maximum of 252 with higher scores indicating higher behavioral challenges.
Trauma Related Symptoms | Assessed at Baseline, 12-weeks post baseline, and at a 3-month follow-up
  Measured by the Child and Adolescent Trauma Screen. The CATS contains 15 items measuring traumatic events, 20 items measuring DSM-5 PTSD symptoms, and 5 items measuring psychosocial functioning, with a range of 0-48 and higher scores indicating greater symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rosmary Ros-Demarize, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Rutledge Tower, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No